CLINICAL TRIAL: NCT02142894
Title: Evaluation of the 4th Generation QuantiFERON-TB Test (CST001) for the Detection of Tuberculosis Infection
Brief Title: Evaluation of the QuantiFERON-TB Test.
Status: Completed | Type: Observational
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CST001_USA1
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; TB
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Symptomatic: Patients with bacteriologically confirmed and untreated TB disease tested with CST001 assay.
  Interventions: Device: CST001

INTERVENTIONS:
Device: CST001

SUMMARY:
To compare the results of the investigational test to the currently approved QuantiFERON-TB Gold In-Tube test.

DETAILED DESCRIPTION:
The objective of the study was to enroll patients who have clinical signs/symptoms strongly indicating TB and who are receiving of have to start the treatment for active TB, and test the variants of the CST001 assay to support the evaluation of clinical sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms consistent with a high probability of having TB disease
* Receiving, or are likely to receive, therapy for active TB
* Confirmed tuberculosis by either AFB smear and culture testing, or Nucleic Acid Amplification methods and culture testing.
* Between 18 and 70 years of age.

Exclusion Criteria:

* Taken therapy for active TB or latent TB for more than 14 days
* Culture confirmation of M. tuberculosis not obtained

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bacteriologically confirmed and untreated TB disease.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2014-05-27 (Actual); Primary Completion 2016-03-28 (Actual); Study Completion 2016-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Jones, MD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Background] QuantiFERON - TB Gold Package Insert (Doc. No. US05990301L). March 2013. Cellestis Inc.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 33 subjects were enrolled.
Groups:
- Symptomatic: Patients with bacteriologically confirmed and untreated TB disease tested with CST001 assay.
  CST001
Period: Overall Study
Arm/Group | Symptomatic
Started | 33
Completed | 25
Not Completed | 8
Not completed — Protocol Violation | 8

BASELINE CHARACTERISTICS:
Arm/Group | Symptomatic
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 21
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Signs/Symptoms Indicating TB With a Positive CST001 Assay Result as an Indication of Clinical Sensitivity
Description: To evaluate the clinical sensitivity of the CST001 assay in patients who have clinical signs/symptoms strongly indicating TB disease and who are receiving or have to start treatment for active TB, and whom Mycobacterium tuberculosis (MTB) is confirmed by bacteriological culture. Patients included in the testing either had a positive acid-fast bacillus (AFB) smear of have MTB in a specimen detected by nucleic acid amplification (NAA) of MTB complex Polymerase Chain Reaction (PCR), and who have received treatment for no more than 14 days upon enrollment.
Time Frame: At time of enrollment
Measure: Count of Participants; unit: Participants
Groups:
- Symptomatic: Evaluation of clinical sensitivity of the CST001 assay in patients who have clinical signs/symptoms indicating TB disease.
Arm/Group | Symptomatic
Number analyzed (Participants) | 33
Participants | 29
Statistical Analysis 1: Comparison: Symptomatic; Test type: Equivalence — The results are analyzed in a 2x2 contingency table with 95%CI; 2 x 2 contingency table = 87.9, 95% CI 2-sided [72.7 to 95.2]

ADVERSE EVENTS:
Time Frame: From 27th May 2014 to 28th Mar 2016.
Arm/Group | Symptomatic
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No